CLINICAL TRIAL: NCT04843228
Title: Combined Cognitive Bias Modification for Perfectionism and Intolerance to Uncertainty: A Randomized Controlled Trial
Brief Title: Cognitive Bias Modification for Perfectionism and Intolerance to Uncertainty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Kübra Tör, MA, Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 13630784
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Perfectionism; Intolerance to Uncertainty
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Condition 1: Cognitive Bias Modification for active group
  Condition 2: Cognitive Bias Modification for control group
Who Masked: Participant, Care Provider
Masking Description: Participants will be blinded to their assigned condition. They will have ID numbers created by random.org which will allow the care provider to be blinded to the assigned conditions of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Cognitive Bias Modification Group (Experimental): This group of participants will receive 4 sessions of CBM targeting their interpretation biases for perfectionism and intolerance to uncertainty.
  Interventions: Behavioral: Cognitive Bias Modification
- Placebo-Control Cognitive Bias Modification Group (Placebo Comparator): This group of participants will receive 4 sessions of inactive CBM.
  Interventions: Behavioral: Cognitive Bias Modification for Control Group

INTERVENTIONS:
Behavioral: Cognitive Bias Modification — There will be four sessions of CBM. Each session will consist of two different part. The first part of the intervention will be the training based on the ambiguous scenario paradigm for perfectionism developed by Dodd (2019). Participants will need to complete word fragments in the last part of the scenario to resolve the ambiguity of the scenario. Then, a comprehension question will be presented to them to underscore the interpretation condition. Feedback will be given after each question. For the second part of the intervention aimed to intervene intolerance to uncertainty, word sentence association paradigm for intolerance to uncertainty developed by Oglesby (2017) will be used. In this intervention, participants will be asked to judge the relatedness of words and sentences which will be presented to them. Feedback will be given after each word-sentence.
  Arms: Active Cognitive Bias Modification Group
Behavioral: Cognitive Bias Modification for Control Group — For the first part of the intervention, the control group will be presented with the same procedures as the active group; however, feedbacks will be given to resolve the scenarios in a neutral way. When it comes to the second part of the intervention, different word-sentence pairings will be presented to the control group.
  Arms: Placebo-Control Cognitive Bias Modification Group

SUMMARY:
This study will examine the impact of cognitive bias modification (CBM) on perfectionism and intolerance to uncertainty. Undergraduate students will be recruited and randomly assigned to either experimental or placebo-control groups. Each group will attend four sessions of CBM over four weeks.

DETAILED DESCRIPTION:
Background. Cognitive bias modification (CBM) is an intervention aiming to systematically change the biases in cognitive processing using experimental paradigms. CBM was found effective with a variety of disorders and transdiagnostic variables. Although there are few studies focusing on transdiagnostic variables like perfectionism and intolerance to uncertainty, further research needs to be done for the generalizability of these results. It was aimed in this study to test the effectiveness of CBM for perfectionism and intolerance to uncertainty with a sample of undergraduate students in Turkey.

Sample size was determined using G*power for a medium to large effect size based on previous studies and it was planned to include 28 undergraduate students who have a score of >70.5 in the Brief Symptom Measure in the study. Participants will get either 3-course credits or a 100 TL bookstore gift card for their full participation. After getting informed consent from participants, they will be randomized to either active or control condition. Participants will be blind to their intervention condition. Following randomization, baseline measurements will be collected. After the baseline measures were collected, links for interventions will be e-mailed to the participants according to their assigned group. Participants will get an email including the link for the study every week. Interpretation bias scores of participants for perfectionism and intolerance to uncertainty will be collected before the first intervention session and after the last intervention session. These sessions will last approximately 25 min. Participants will attend the session without an assessment in the second and third week and these sessions will last approximately 15 min. After four sessions, post-tests will be sent to the participants. Questionnaires will also be collected one month after the intervention was done.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* Have a score of >70.5 in Brief Symptom Measure
* Being an undergraduate student
* Fluent in Turkish
* Access to the internet by computer

Exclusion Criteria:

* Having any psychiatric disorder
* Receiving a psychiatric/psychological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change in Brief Symptom Measure | Weeks 0, 4, 8
  Psychiatric symptomatology will be assessed with Brief Symptom Measure consists of 25 items scored 1-7. Greater score means greater severity.

SECONDARY OUTCOMES:
Change in Interpretation bias for perfectionism | Weeks 0, 4
  Participants will read ten scenarios and rate the relatedness of four sentences for each scenario.
Change in Interpretation bias for intolerance to uncertainty | Weeks 0, 4
  Participants will judge the relatedness of word-sentence pairings. 40 pairings will be presented and each participant will have a score between 0 and 1. A score closer to 0 indicates severity of interpretation bias for intolerance to uncertainty.
Change in Frost Multidimensional Perfectionism Scale | Weeks 0, 4, 8
  Self-report questionnaire of perfectionism consists of 35 items on a 5-point scale. Higher score means greater perfectionism.
Change in Intolerance of Uncertainty Scale | Weeks 0, 4, 8
  Self-report questionnaire of intolerance to uncertainty consists of 26 items on a 5-point scale. Higher score means greater intolerance to uncertainty.
Change in Cognitive-Behavioral Avoidance Scale | Weeks 0, 4, 8
  Self-report questionnaire of cognitive-behavioral avoidance consists of 31 items on a 5-point scale. Higher score means greater cognitive-behavioral avoidance.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Lowell, Lowell, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No